CLINICAL TRIAL: NCT03370744
Title: Prediction of Cognitive Decline by Neuroimaging Techniques and the Application in Diagnosis and Treatment of Preclinical AD (Sino Longitudinal Study on Cognitive Decline, SILCODE)
Brief Title: Prediction of Cognitive Decline by Neuroimaging Techniques and the Application in Diagnosis and Treatment of Preclinical AD
Status: Completed | Type: Observational
Sponsor: XuanwuH 2 (Other)
Responsible Party: Sponsor-Investigator, XuanwuH 2, Director of Neurology, Professor, Xuanwu Hospital, Beijing
Organization: Xuanwu Hospital, Beijing (Other)
Other Study IDs: hanying4
Record Dates: First submitted 2017-11-15; First posted 2017-12-12 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Subjective Cognitive Decline; Preclinical Alzheimer's Disease
Keywords: subjective cognitive decline; brain network; multi-modality; magnetic resonance imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Subjective cognitive decline, SCD: The inclusion criteria for SCD are as following: (1) presence of self-perceived continuous cognitive decline compared to previous normal status and unrelated to an acute event; and (2) failure to meet the following criteria for MCI.
  Interventions: Diagnostic Test: Neuropsychological scale
- Normal control, NC: NC are individuals who have no self-report persistent decline in cognitive capacity, and with neither worry nor concern about their cognition. Without measurable cognitive impairment according to results of standard assessments.
  Interventions: Diagnostic Test: Neuropsychological scale
- Mild cognitive impairment, MCI: MCI are defined by an actuarial neuropsychological method proposed by Jak and Bondi. Participants are considered to have MCI if any one of the following three criteria are met with a total Clinical Dementia Rating (CDR) score of 0.5 as well as failure to meet the criteria for dementia: (1) having impaired scores (defined as >1 SD below the age-corrected normative mean) on both measures within at least one cognitive domain (i.e., memory, language, or speed/executive function); (2) having impaired scores in each of the three cognitive domains sampled; (3) the Functional Activities Questionnaire (FAQ) ≥9.
  Interventions: Diagnostic Test: Neuropsychological scale
- Alzheimer's disease, AD: The diagnosis of AD syndrome is based on the diagnostic guidelines for dementia due to AD delivered by the National Institute on Aging-Alzheimer's Association workgroups (NIA-AA) with a total CDR score of 1.
  Interventions: Diagnostic Test: Neuropsychological scale
- Subjective Cognitive Decline plus, SCD-plus: The inclusion criteria for SCD-plus are as following: (1) presence of self-perceived continuous cognitive decline compared to previous normal status and unrelated to an acute event; and (2) concerns (worries) associated with memory complaint; and (3) failure to meet the following criteria for MCI.
  Interventions: Diagnostic Test: Neuropsychological scale

INTERVENTIONS:
Diagnostic Test: Neuropsychological scale — Neuropsychological scale, including mini-mental state examination (MMSE), Montreal cognitive assessment (MoCA), clinical dementia rating scales (CDR) and so on

SUMMARY:
This study is affiliated to Sino Longitudinal Study on Cognitive Decline, SILCODE. To establish models of normal and pathological cognitive aging.To collect the longitudinal data of SCD population, to study the dynamic changes of brain networks so as to explore the progressive mechanisms of AD on brain networks and to construct a high-precision multi-modal model for early diagnosis.

DETAILED DESCRIPTION:
This study is affiliated to Sino Longitudinal Study on Cognitive Decline, SILCODE. Alzheimer's disease (AD) is the most common cause of dementia, which severely injures multiple domains of cognitive functions in the aging people, bringing heavy burden to the society and families. Studying the cognitive brain damage mechanism of subjective cognitive decline (SCD), the preclinical stage of AD, would provide great opportunities for understanding the pathogenesis of AD and clinical value for early diagnosis and intervention in AD. The project intends to utilize amyloid-PET and FDG-PET for screening and then employ the comprehensive neuropsychological examination combined with multi-modal MRI neuroimaging techniques to study the brain functions and structures of the normal aging and SCD. The imaging data would be analyzed from several levels, including the cognitive dimensions, brain activation patterns, and especially functional and structural networks to establish the models of normal and pathological cognitive aging, which mainly be modulated by frontal-parietal control system. We aim to establish models of normal and pathological cognitive aging. Furthermore, the longitudinal data of SCD population would be collected to study the dynamic changes of brain networks so as to explore the progressive mechanisms of AD on brain networks and to construct a high-precision multi-modal model for early diagnosis

ELIGIBILITY:
1. NC Inclusion Criteria:

1. Older than 60, right handedness, Han nationality;
2. Have no cognitive decline complains, with neither worry nor concern about their cognition;
3. Scores of standardized neuropsychological tests scale adjusted for age, sex and education are in normal range;
4. Physical examination is negative;
5. Review medical history and family history is negative, accessory examination don't show disease could cause cognitive decline;
6. Could cooperate collection of multi-modal magnetic resonance imaging, once a year, for continueously five years.

2. SCD Inclusion Criteria:

1. Presence of self-perceived continuous cognitive decline compared to previous normal status and unrelated to an acute event;
2. Failure to meet the following criteria for MCI.

3.SCD-plus Inclusion Criteria:

1. Presence of self-perceived continuous cognitive decline compared to previous normal status and unrelated to an acute event;
2. Concerns (worries) associated with memory complaint;
3. Failure to meet the following criteria for MCI.

3. MCI Inclusion Criteria:

1. Clinical Dementia Rating (CDR) score of 0.5 as well as failure to meet the criteria for dementia
2. Having impaired scores (defined as >1 SD below the age-corrected normative mean) on both measures within at least one cognitive domain (i.e., memory, language, or speed/executive function);
3. Having impaired scores in each of the three cognitive domains sampled;
4. the Functional Activities Questionnaire (FAQ) ≥9.

4. AD Inclusion Criteria The diagnosis of AD syndrome is based on the diagnostic guidelines for dementia due to AD delivered by the National Institute on Aging-Alzheimer's Association workgroups (NIA-AA)with a total CDR score of 1.

Exclusion Criteria:

1. Claustrophobia, with metals in the body that cannot be examined by MRI, including metal dentures or other contraindications for examination;
2. Left handedness or ambidextrality.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers recrewed from communities, and signed up with informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The altered volume pattern in SCD/SCD-plus with progression. | 5 years
  1. Global grey matter volume change of brain in µm3
  2. Regional gray matter volume change of brain in µm3
  3. Cerebral cortex thickness change of brain in µm
The altered DTI pattern in SCD/SCD-plus with progression. | 5 years
  1. Regional fractional anisotropy (FA), measured by diffusion tensor imaging (DTI).
  2. Regional mean diffusivity (MD), measured by DTI.
  3. Regional radial diffusivity (RD), measured by DTI.
  4. Regional axial diffusivity (AxD), measured by DTI.
The altered functional MRI pattern in SCD/SCD-plus with progression. | 5 years
  Resting state functional MRI blood-oxygen-level-dependent (fMRI BOLD) signal.
The altered FDG-PET pattern in SCD/SCD-plus with progression. | 5 years
  Global SUVR change of brain of FDG-PET in kBq/ml/MBq/kg.
The altered AV45-PET pattern in SCD/SCD-plus with progression. | 5 years
  Global SUVR change of brain of AV45-PET in kBq/ml/MBq/kg.
Genotype of SCD/SCD-plus with progression. | 5 years
  ApoE genotype by blood test.
AD7c-NTP level of SCD/SCD-plus with progression. | 5 years
  AD7c-NTP level by urine tests.
Gut microbiota of SCD/SCD-plus with progression. | 5 years
  Gut microbiota level by 16s rDNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Ying Han, Doctor, Study Chair — Xuanwu Hospitial Capital Medical University
Locations (1):
- Department of Neurolgy,Xuanwu Hospital of Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen HJ, Zhang M, Wei M, Yu X, Wang Y, Yang J, Li R, Zhao W, Wang X, Zhang S, Wang K, Bai T, Huo Y, Huang W, Dai Z, Ma G, Han Y, Chen G, Shu N. Amyloid pathology related to aberrant structure-function coupling of brain networks in Alzheimer's disease: insights from [18F]-florbetapir PET imaging. Eur J Nucl Med Mol Imaging. 2025 Jul;52(8):2929-2940. doi: 10.1007/s00259-025-07172-8. Epub 2025 Mar 7. PMID 40053120
- [Derived] Zhao C, Li T, Hao S, Zhao L, Han Y, Cai Y. Dysregulation of the molecular clock by blood-borne factors in Alzheimer's disease patients. J Neurol. 2025 Jan 15;272(2):121. doi: 10.1007/s00415-024-12824-0. PMID 39812690
- [Derived] Yu X, Zhang Y, Cai Y, Rong N, Li R, Shi R, Wei M, Jiang J, Han Y. Asymmetrical patterns of beta-amyloid deposition and cognitive changes in Alzheimer's disease: the SILCODE study. Cereb Cortex. 2024 Dec 3;34(12):bhae485. doi: 10.1093/cercor/bhae485. PMID 39710611
- [Derived] Wang L, Xu H, Wang M, Brendel M, Rominger A, Shi K, Han Y, Jiang J. A metabolism-functional connectome sparse coupling method to reveal imaging markers for Alzheimer's disease based on simultaneous PET/MRI scans. Hum Brain Mapp. 2023 Dec 1;44(17):6020-6030. doi: 10.1002/hbm.26493. Epub 2023 Sep 23. PMID 37740923
- [Derived] Wang T, Yao Y, Han C, Li T, Du W, Xue J, Han Y, Cai Y. MCP-1 levels in astrocyte-derived exosomes are changed in preclinical stage of Alzheimer's disease. Front Neurol. 2023 Mar 20;14:1119298. doi: 10.3389/fneur.2023.1119298. eCollection 2023. PMID 37021284
- [Derived] Wang T, Wang X, Yao Y, Zhao C, Yang C, Han Y, Cai Y. Association of plasma apolipoproteins and levels of inflammation-related factors with different stages of Alzheimer's disease: a cross-sectional study. BMJ Open. 2022 Apr 6;12(4):e054347. doi: 10.1136/bmjopen-2021-054347. PMID 35387811
- [Derived] Sheng C, Yang K, He B, Du W, Cai Y, Han Y. Combination of gut microbiota and plasma amyloid-beta as a potential index for identifying preclinical Alzheimer's disease: a cross-sectional analysis from the SILCODE study. Alzheimers Res Ther. 2022 Feb 14;14(1):35. doi: 10.1186/s13195-022-00977-x. PMID 35164860
- [Derived] Ding C, Du W, Zhang Q, Wang L, Han Y, Jiang J. Coupling relationship between glucose and oxygen metabolisms to differentiate preclinical Alzheimer's disease and normal individuals. Hum Brain Mapp. 2021 Oct 15;42(15):5051-5062. doi: 10.1002/hbm.25599. Epub 2021 Jul 22. PMID 34291850
- [Derived] Dong QY, Li TR, Jiang XY, Wang XN, Han Y, Jiang JH. Glucose metabolism in the right middle temporal gyrus could be a potential biomarker for subjective cognitive decline: a study of a Han population. Alzheimers Res Ther. 2021 Apr 7;13(1):74. doi: 10.1186/s13195-021-00811-w. PMID 33827675
- [Derived] Sheng C, Sun Y, Wang M, Wang X, Liu Y, Pang D, Liu J, Bi X, Du W, Zhao M, Li Y, Li X, Jiang J, Han Y. Combining Visual Rating Scales for Medial Temporal Lobe Atrophy and Posterior Atrophy to Identify Amnestic Mild Cognitive Impairment from Cognitively Normal Older Adults: Evidence Based on Two Cohorts. J Alzheimers Dis. 2020;77(1):323-337. doi: 10.3233/JAD-200016. PMID 32716355
- [Derived] Li X, Wang X, Su L, Hu X, Han Y. Sino Longitudinal Study on Cognitive Decline (SILCODE): protocol for a Chinese longitudinal observational study to develop risk prediction models of conversion to mild cognitive impairment in individuals with subjective cognitive decline. BMJ Open. 2019 Jul 26;9(7):e028188. doi: 10.1136/bmjopen-2018-028188. PMID 31350244
- [Derived] Sun Y, Wang X, Wang Y, Dong H, Lu J, Scheininger T, Ewers M, Jessen F, Zuo XN, Han Y. Anxiety correlates with cortical surface area in subjective cognitive decline: APOE epsilon4 carriers versus APOE epsilon4 non-carriers. Alzheimers Res Ther. 2019 Jun 3;11(1):50. doi: 10.1186/s13195-019-0505-0. PMID 31159873